CLINICAL TRIAL: NCT02254694
Title: The Influence of High Heeled Shoes on the Sagittal Balance of the Spine and Whole Body
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: SNCTP000000049
Record Dates: First submitted 2014-09-18; First posted 2014-10-02 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Back Pain
Keywords: sagittal balance; posture; lumbar lordosis; high heeled shoes
MeSH Terms: conditions — Back Pain; Lordosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- high heeled shoes (Experimental): see detailed description
  Interventions: Other: high heeled shoes

INTERVENTIONS:
Other: high heeled shoes — see detailed study description

SUMMARY:
The purpose of this study is to investigate the influence of high heeled shoes on the sagittal balance of the spine and the whole body.

The investigators hypothesize that wearing high heeled shoes leads to a hyperlordosis of the cervical spine, a decrease of thoracic kyphosis, hyperlordosis of the lumbar spine and a posterior tilt of the pelvis resulting in a posterior shift of the body's center of gravity. This would be an explanation for the increased prevalence of back pain in individuals frequently wearing high heels.

In order to assess these changes, differences in the two following outcome parameters will be measured on a standing lateral EOS-radiograph of the whole body - barefoot and with high heeled shoes: spino-sacral angle (primary) and meatus plumb line (secondary) .

DETAILED DESCRIPTION:
Female volunteers (age ≥ 21 years) that are not frequent user of high heeled shoes (i.e. not longer than 6 hours/month with heels > 3 cm) will be included. Exclusion criteria are osseous metastases, missing written informed consent, cognitive inability to consent on their own, and pregnancy. Based on own preliminary studies, a sample size of 19 (+3 to anticipate drop outs) patients is aimed for.

After obtaining informed consent, the participants will be interviewed with special regard to their age, gender, height, weight, shoe size, past medical history, occupational and recreational activities, and duration and frequency of wearing high heeled shoes.

A clinical examination of the spine and pelvis will be performed as well as a pregnancy urine test.

Standing lateral EOS-radiographs (http://www.eos-imaging.com/) of the whole body will be taken - once barefoot and once with high heeled shoes (heel height 9 cm).

All data acquisition is going to be performed during a single session, participants will not be followed up.

The following parameters will be assessed on the radiographs: presence and number of (healed) fractures, osseous metastases, sagittal C7 plumb line, meatus plumb line, cervical lordosis, thoracic kyphosis, lumbar lordosis, spino- sacral angle as described by Roussouly et al. (2006), pelvic incidence, pelvic tilt.

For statistical analysis, all data will be collected in a statistic software file (SPSS. 21.0, SPSS Inc, Chicago, Illinois). After testing for normal distribution, these differences in means of the primary and secondary outcome parameters between the barefoot and the high heeled radiograph will be assessed using a paired Student's T-test or non-parametric tests. The level of significance is p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* not frequent user of high heeled shoes (i.e. not longer than 6 hours/month with heels > 3 cm)

Exclusion Criteria:

* osseous metastases
* missing written informed consent
* cognitive inability to consent on their own
* pregnancy

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2014-09; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
spino-sacral angle | 1 day
  "spino-sacral angle" measured on the lateral EOS-radiograph of the whole body as described in: "Classification of the normal variation in the sagittal alignment of the human lumbar spine and pelvis in the standing position." Roussouly P, Gollogly S, Berthonnaud E, Dimnet J. Spine (Phila Pa 1976). 2005 Feb 1;30(3):346-53.

SECONDARY OUTCOMES:
meatus plumb line | 1 day
  plumb line from the meatus acusticus in relation to the calcaneal tuberosity on the lateral radiograph of the whole body

CONTACTS AND LOCATIONS:
Overall Officials: Clément ML Werner, MD, Prof, Principal Investigator — University of Zurich, Klinik für Unfallchirurgie
Locations (1):
- Klinik für Unfallchirurgie, University Hospital Zurich, Zurich, Canton of Zurich, Switzerland

REFERENCES:
- [Result] Opila KA, Wagner SS, Schiowitz S, Chen J. Postural alignment in barefoot and high-heeled stance. Spine (Phila Pa 1976). 1988 May;13(5):542-7. doi: 10.1097/00007632-198805000-00018. PMID 3187700